CLINICAL TRIAL: NCT00259519
Title: Effects of Intentional Delivery After Preterm and Prelabor Rupture of Membranes Between 32 and 35 Weeks of Gestation: A Multicentre Randomized and Controlled Trial
Brief Title: Safety and Efficacy Study of Intentional Delivery in Women With Preterm and Prelabour Rupture of the Membranes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The DSMB supported termination of the trial due to slow recruitment.
Sponsor: University of Alberta (Other)
Collaborators: Stollery Children's Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N041000314
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Fetal Membranes, Premature Rupture
Keywords: premature or preterm birth; chorioamnionitis; neonatal sepsis; labour; Cesarean Section; delivery; length of stay; pregnancy
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Premature Birth; Chorioamnionitis; Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Expectant management
- 2 (Active Comparator): Induction of delivery
  Interventions: Procedure: Induction of delivery

INTERVENTIONS:
Procedure: Induction of delivery — Induction of delivery
  Other Names: immediate delivery
  Arms: 2

SUMMARY:
Two-year multicentre randomized controlled parallel trial to compare intentional delivery and conservative management in pregnant women with preterm and prelabour rupture of membranes between 32 and 35 weeks.

The purpose of this study is to determine whether intentional delivery of women with PPROM between 32 and 35 week's gestation can decrease the overall neonatal morbidity associated with PPROM-related complications without increasing the morbidity associated with a shortened pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women with recent PPROM between 31 weeks + 6 days and 35 weeks + 6 days (estimated gestational age based on an ultrasound examination before 18 weeks of gestation), not in labour 24 hours after admission*, will be considered eligible for the study provided the following inclusion criteria (*For patients transferred from a remote level 2 centre to one of the participating sites within the first hours after PPROM, the onset of the 24-hour screening period will be the time of admission in the centre of origin. Patients in Group A will be given their first dose of antenatal steroids before the transfer)
* Single and otherwise uncomplicated pregnancy
* Recent history (less than 48 hours) of leaking with the two followings within 24 hours after primary medical assessment: Documentation of fluid from the vagina and Positive Fern test, or positive Nitrazine test, or Positive ACTIM PROM test
* Antenatal steroids course initiated after the rupture for women with PPROM between 31 + 6 and 33 + 6 weeks
* Normal fetal heart rate trace using an external ultrasound transducer
* Written informed consent obtained before inclusion and randomization

Exclusion Criteria:

* Multiple pregnancy
* HIV positive mother
* Active HSV cervical lesions
* Major fetal anomaly on ultrasound examination performed after admission
* Intrauterine growth restriction estimated on ultrasound below the 5th percentile or preeclampsia
* Placenta abruption present at the time of the diagnosis of PPROM or occurring within the first 24 hours after rupture
* Clinical chorioamnionitis existing before or at the time of the diagnosis of PPROM or developing within the first 24 hours after rupture
* Non-reassuring fetal testing present at the time of the diagnosis of PPROM or occurring within the first 24 hours after the rupture. It implies that expected criteria for standard fetal assessment parameters have not been met, including the Non-Stress test and the Biophysical profile Score. This will be diagnosed at the discretion of the attending physician.
* More generally, any maternal or fetal reason for an immediate delivery, either existing at admission or occurring within the 24 hours after admission.
* Mother refusal or inability to provide consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Length of Stay in hospital | time between birth and readiness for discharge

SECONDARY OUTCOMES:
MAIN Score (Morbidity Assessment Index for Newborns) | From birth to discharge
Early Onset Neonatal Sepsis | from birth to discharge
Clinical and Histological Chorioamnionitis | from birth to discharge
Antepartum Length of stay | From diagnosis to delivery
C-Section | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lacaze-Masmonteil, MD, PhD, Principal Investigator — University of Alberta; Radha Chari, MD,FRCPC, Principal Investigator — University of Alberta- Department of Gynecology and Obstetrics
Locations (11):
- Canada (11):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Caritas - Misericordia Hospital, Edmonton, Alberta
  - BC Women's Hospital and Health Centre, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Women's Hospital, Winnipeg, Manitoba
  - Saint-Joseph Health Care, London, Ontario
  - Sainte-Justine Hospital, Montreal, Quebec
  - Laval University Hospital, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan